CLINICAL TRIAL: NCT01242267
Title: A Phase I/II Study of Escalating Doses of Thalidomide in Conjunction With Bortezomib and HIgh Dose Melphalan as a Conditioning Regimen for Autologous Peripheral Blood Stem Cell Transplantation in Patients With Advanced Multiple Myeloma
Brief Title: Escalating Doses of Thalidomide in Conjunction With Bortezomib and HIgh Dose Melphalan for BSCT
Acronym: Thal/Mel/Vel
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hackensack Meridian Health (Other)
Collaborators: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRO00001215
Record Dates: First submitted 2010-11-15; First posted 2010-11-16 (Estimated); Results first posted 2023-01-03 (Actual); Last update posted 2023-01-03 (Actual); Status verified 2022-12

CONDITIONS: Multiple Myeloma
Keywords: multiple myeloma; transplant; Multiple myeloma patients undergoing transplant
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Phase 1 (Experimental): Phase 1 including Thalidomide Dose Levels of 600, 800, 1000 mg. Three patients will be entered at each dose level sequentially with a maximum of six patients enrolled at the highest dose level that defines dose-limiting toxicity. The starting dose will be 600mg/d x 5 days (dose level 1) given on days -5 to -1 before transplantation. Doses will be escalated in sequential order as listed below through cohorts of patients.
  Interventions: Drug: Thalidomide+Melphalan +Bortezomib+stem cell transplant
- Phase 2 (Experimental): Phase 2 Thalidomide Dose Level of 1000 mg. The maximum dose to be tested is 1000mg. When the MTD is defined, an additional 40 patients will be enrolled at this level. The first 3 patients of this cohort of 40 patients will be assessed for DLT (2 of 6 patients experiencing DLT at this dose will require dose-de-escalation as described above, and the phase II portion of the study re-initiated at the newly defined MTD).
  Interventions: Drug: Thalidomide+Melphalan +Bortezomib+stem cell transplant

INTERVENTIONS:
Drug: Thalidomide+Melphalan +Bortezomib+stem cell transplant — Five days prior to transplant, the patient starts thalidomide. Dose range will be from 600mg for 5 days, to 1000mg for 5 days. Thalidomide dose is increased after groups of 3 to 6 patients have been treated. 4 days before the transplant and again on the day before the transplant the patient will be given bortezomib (VELCADE) intravenously at a dose of 1.6 mg/m2 (mg/m2 means that the dose will be calculated based on the patient's height and weight). 2 days before transplant the patient will be given melphalan 200 mg/m2 intravenously. Dexamethasone is given before the VELCADE and the melphalan.

SUMMARY:
The primary objective of this study is to:

• Determine the maximum tolerated dose of thalidomide used in conjunction with dose-intense melphalan, bortezomib and autologous (syngeneic) HSC support in the salvage therapy of patients who failed a prior treatment with dose-intense melphalan

The secondary objectives of this study are to:

* Determine the toxicities resulting from administration of combinations of thalidomide, bortezomib and melphalan
* Determine the complete response (CR) and very good partial response (VgPR) rate in patients undergoing ASCT using thalidomide, bortezomib and melphalan
* Evaluate the treatment-free interval after treatment with the combination of thalidomide, bortezomib and melphalan

DETAILED DESCRIPTION:
VELCADE™ (bortezomib) for Injection is a small molecule proteasome inhibitor developed by Millennium Pharmaceuticals, Inc., (Millennium) as a novel agent to treat human malignancies. VELCADE is currently approved by the United States Food and Drug Administration (US FDA) and it is registered in Europe for the treatment of multiple myeloma patients who have received at least one prior therapy.

By inhibiting a single molecular target, the proteasome, bortezomib affects multiple signaling pathways. The anti-neoplastic effect of bortezomib likely involves several distinct mechanisms, including inhibition of cell growth and survival pathways, induction of apoptosis, and inhibition of expression of genes that control cellular adhesion, migration and angiogenesis. Thus, the mechanisms by which bortezomib elicits its antitumor activity may vary among tumor types, and the extent to which each affected pathway is critical to the inhibition of tumor growth could also differ. Bortezomib has a novel pattern of cytotoxicity in National Cancer Institute (NCI) in vitro and in vivo assays (Adams et al., 1999). In addition, bortezomib has cytotoxic activity in a variety of xenograft tumor models, both as a single agent and in combination with chemotherapy and radiation (Steiner et al., 2001; Teicher et al., 1999; Cusack et al., 2001; LeBlanc et al., 2002; Pink et al., 2002). Notably, bortezomib induces apoptosis in cells that over express bcl-2, a genetic trait that confers unregulated growth and resistance to conventional chemotherapeutics (McConkey et al., 1999).

Bortezomib is thought to be efficacious in multiple myeloma via its inhibition of nuclear factor κB (NF-κB) activation, its attenuation of interleukin-6 (IL-6)-mediated cell growth, a direct apoptotic effect, and possibly anti-angiogenic and other effects.

ELIGIBILITY:
Inclusion Criteria:

* Each patient must meet all of the following inclusion criteria to be enrolled in the study:
* Voluntary written informed consent before performance of any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the subject at any time without prejudice to future medical care
* Female subject is either post-menopausal or surgically sterilized or willing to use an acceptable method of birth control as described in the S.T.E.P.S program. Participation in the program is required.
* Male subject agrees to use an acceptable method for contraception for the duration of the study as described in the S.T.E.P.S program. Participation in the program is required.
* Confirmed diagnosis of multiple myeloma, or plasma cell leukemia.
* Show progression of disease after a previous dose-intense cycle of melphalan, or less than a complete response after a prior cycle of dose-intense melphalan. Patients may have received more than on prior autologous transplant with high-dose melphalan.
* May have received intervening therapies after disease progression after dose-intense melphalan and before enrollment in this protocol.
* Recovery from complications of salvage therapy, if administered.
* Age: ≥18 yrs but <76 yrs at the time of melphalan administration.
* Gender: There is no gender restriction.
* Availability of >2x106 autologous peripheral blood CD34+ cells/kg or a syngeneic donor meeting eligibility criteria for syngeneic donation.

  1. Syngeneic transplantation is preferred.

Exclusion Criteria:

* Patients meeting any of the following exclusion criteria are not to be enrolled in the study.
* Cytotoxic chemotherapy or radiotherapy within 21 days of initiating treatment in this study.
* Prior dose-intense therapy within 56 days of initiating treatment in this study.
* Uncontrolled bacterial, viral, fungal or parasitic infections .
* Uncontrolled CNS metastases.
* Known amyloid deposition in heart.
* Organ dysfunction:

LVEF <40% or cardiac failure not responsive to therapy. DLCO <50% of predicted and/or receiving supplementary continuous oxygen. Evidence of hepatic synthetic dysfunction, or total bilirubin >2x or AST >3x ULN.

Measured creatinine clearance <20 ml/min. Sensory peripheral neuropathy grade 4 within 14 days of enrollment.

* Karnofsky score <70% unless as a result of bone disease directly caused by myeloma.
* Life expectancy limited by another co-morbid illness.
* Diagnosed or treated for another malignancy within 2 years of enrollment, with the exception of complete resection of basal cell carcinoma or squamous cell carcinoma of the skin, an in situ malignancy, or low-risk prostate cancer after curative therapy
* Female subject is pregnant or breast-feeding (women) or unwilling to use acceptable birth control methods (men or women) for twelve months after treatment or unwilling to participate in the S.T.E.P.S program.
* Documented hypersensitivity to melphalan, thalidomide or to bortezomib, boron or mannitol or any components of the formulation
* Patients unable or unwilling to provide consent
* Myocardial infarction within 6 months prior to enrollment or has New York Heart Association (NYHA) Class III or IV heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities. Prior to study entry, any ECG abnormality at screening has to be documented by the investigator as not medically relevant.
* Patient has received other investigational drugs with 14 days before enrollment
* Serious medical or psychiatric illness likely to interfere with participation in this clinical study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2010-05-11 (Actual); Primary Completion 2016-01-20 (Actual); Study Completion 2016-01-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott D Rowley, MD, Principal Investigator — John Theurer Cancer Center at Hackensack Univ Medical Center
Locations (1):
- John Theurer Cancer Center at Hackensack University Medical Center, Hackensack, New Jersey, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase I - Thalidomide Dose Level 600 mg: Phase I - Thalidomide Dose Level 600 mg
- Phase I - Thalidomide Dose Level 800 mg: Phase I - Thalidomide Dose Level 800 mg
- Phase I - Thalidomide Dose Level 1000 mg: Phase I - Thalidomide Dose Level 1000 mg
- Phase 2: Phase 2 Thalidomide Dose Level 1000 mg
Period: Overall Study
Arm/Group | Phase I - Thalidomide Dose Level 600 mg | Phase I - Thalidomide Dose Level 800 mg | Phase I - Thalidomide Dose Level 1000 mg | Phase 2
Started | 3 | 3 | 3 | 20
Completed | 3 | 3 | 3 | 20
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Phase II: Phase II Thalidomide Dose Level 1000 mg
- Total: Total of all reporting groups
Arm/Group | Phase I - Thalidomide Dose Level 600 mg | Phase I - Thalidomide Dose Level 800 mg | Phase I - Thalidomide Dose Level 1000 mg | Phase II | Total
Number analyzed (Participants) | 3 | 3 | 3 | 20 | 29
Age, Customized [Median (Full Range); unit: years]
  Range | 66 [58 to 69] | 59 [50 to 70] | 52 [52 to 64] | 55 [40 to 70] | 56 [40 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3 | 9 | 15
  Male | 2 | 1 | 0 | 11 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 1 | 2
  Not Hispanic or Latino | 3 | 3 | 2 | 19 | 27
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 4 | 5
  White | 2 | 3 | 2 | 14 | 21
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 2 | 2
Region of Enrollment [Number; unit: participants]
  United States | 3 | 3 | 3 | 20 | 29

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose of Thalidomide
Description: Maximum tolerated dose of thalidomide used in conjunction with dose-intense melphalan, bortezomib and autologous (syngeneic) HSC support in the salvage therapy of patients who failed a prior treatment with dose-intense melphalan
Time Frame: Dose escalation will be based on the assessment of tolerability determined after the last patient of each cohort reaches day +21.
Measure: Number; unit: mg
Groups:
- Phase 1: Phase 1 Dose Level 600, 800, 1000 mg of Thalidomide
- Phase 2: Phase 2 Dose Level 1000 mg of Thalidomide
Arm/Group | Phase 1 | Phase 2
Number analyzed (Participants) | 9 | 20
mg | 1000 | 1000

2. Secondary Outcome: Complete Response (CR) and Very Good Partial Response (VgPR) Rate
Description: The complete response (CR) and very good partial response (VgPR) rate in patients undergoing ASCT using thalidomide, bortezomib and melphalan
Time Frame: Assessments will be made from Day +28 after transplantation for 3 months and then at 3 month intervals until demonstration of disease progression and initiation of further therapy, an average of 9 months
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I - Thalidomide Dose Level 600 mg | Phase I - Thalidomide Dose Level 800 mg | Phase I - Thalidomide Dose Level 1000 mg | Phase 2
Number analyzed (Participants) | 3 | 3 | 3 | 20
Participants | 0 | 3 | 1 | 13

3. Secondary Outcome: Toxicity Assessment
Description: Assessment of the toxicities resulting from administration of combinations of thalidomide, bortezomib and melphalan
Time Frame: Patients will be hospitalized or in the outpatient transplant facility until engraftment and resolution of serious adverse events, a median of 16 (range, 11-24) days
Measure: Number; unit: Serious Adverse Events
Arm/Group | Phase I - Thalidomide Dose Level 600 mg | Phase I - Thalidomide Dose Level 800 mg | Phase I - Thalidomide Dose Level 1000 mg | Phase 2
Number analyzed (Participants) | 3 | 3 | 3 | 20
Serious Adverse Events | 1 | 0 | 0 | 3

4. Secondary Outcome: Treatment Free Interval/PFS
Description: The treatment-free interval after treatment with the combination of thalidomide, bortezomib and melphalan
Time Frame: PFS was defined as the time from ASCT to disease progression or death from any cause, an average of 9 months
Population: Data no longer available, only manuscript information where PFS reported for single Arm/Group of all participants
Measure: Median (Standard Deviation); unit: months
Groups:
- Phase 1/Phase 2: Assessment of PFS made using the entire cohort
Arm/Group | Phase 1/Phase 2
Number analyzed (Participants) | 29
months | 9.3 (0)

ADVERSE EVENTS:
Description: The limited number of patients limited our ability to analyze groups separately. As a result, all subjects in the Phase I portion were combined to produce a meaningful analysis.
Arm/Group | Phase I - Thalidomide Dose Level 600 mg | Phase I - Thalidomide Dose Level 800 mg | Phase I - Thalidomide Dose Level 1000 mg | Phase 2
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3 | 0/3 | 0/20
Serious Adverse Events (participants affected / at risk) | 1/3 | 0/3 | 0/3 | 3/20
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 3/3 | 20/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I - Thalidomide Dose Level 600 mg (N=3) | Phase I - Thalidomide Dose Level 800 mg (N=3) | Phase I - Thalidomide Dose Level 1000 mg (N=3) | Phase 2 (N=20)
Engraftment Syndrome with GI Invovlement (Blood and lymphatic system disorders) | 1 (1) | NA | NA | 0 (0)
Rheumatoid Arthritis Flare (Immune system disorders) | 0 (0) | NA | NA | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | NA | NA | 1 (1)
Tumor Lysis Syndrome (Metabolism and nutrition disorders) | 0 (0) | NA | NA | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I - Thalidomide Dose Level 600 mg (N=3) | Phase I - Thalidomide Dose Level 800 mg (N=3) | Phase I - Thalidomide Dose Level 1000 mg (N=3) | Phase 2 (N=20)
Hypotension (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulmonary Hypertension (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mild Left Atrial Dilatation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Deep Venous Thrombosis (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Nausea (Gastrointestinal disorders) | 2 (2) | 3 (3) | 2 (2) | 13 (13)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 3 (3) | 1 (1) | 10 (10)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 3 (3)
Anorexia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Mucositis (Gastrointestinal disorders) | 2 (2) | 0 (0) | 2 (2) | 13 (13)
Acid Reflux (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dry Mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal Pain/Cramping (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Odynophagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Dysgeusia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Somnolence (Nervous system disorders) | 3 (3) | 3 (3) | 3 (3) | 7 (7)
Neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 4 (4)
Fatigue (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 5 (5)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Failure to Thrive (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Renail Impairment (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Fluid Overload (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary Hesitancy (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Prostatism (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tumor Lysis Syndrome (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fever (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Febrile Neutropenia (Infections and infestations) | 1 (1) | 1 (1) | 2 (2) | 13 (13)
Febrile Neutropenia (culture-negative) (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 12 (12)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Upper Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Joint Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Joint Effusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Weakness Low Extremity/Generalized (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 7 (7)
Low Extremity Pain/Cramping (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Low Extremity Edema (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Soft Tissue Mass of the Hand (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Breast Discomfort (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes